CLINICAL TRIAL: NCT04667260
Title: Maxillary Sinus Floor Augmentation With a 1:1 Mixture of Autogenous Bone Graft and Symbios Xenograft Granules Compared With Blood Coagulum. A Randomized Controlled Trial
Brief Title: Sinus Floor Augmentation and Graft Compared Sinus Membrane Elevation With Blood Coagulum. A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Thomas Starch-Jensen, Professor, DDS, PhD, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-20180080
Record Dates: First submitted 2020-11-30; First posted 2020-12-14 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Dental Implant Failed
MeSH Terms: interventions — Sinus Floor Augmentation

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Masking Description: Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bone substitue (Placebo Comparator): Bone augmentation with bone substitute
  Interventions: Procedure: Maxillary sinus membrane elevation; Procedure: Maxillary sinus floor augmentation
- Coagulum (Experimental): Bone augmentation with coagulum
  Interventions: Procedure: Maxillary sinus membrane elevation; Procedure: Maxillary sinus floor augmentation

INTERVENTIONS:
Procedure: Maxillary sinus membrane elevation — Maxillary sinus membrane elevation with blood coagulum
  Other Names: Sinus membrane elevation
Procedure: Maxillary sinus floor augmentation — Maxillary sinus floor augmentation with 1:1 autogenous bone graft and deprotinized porcine bone mineral
  Other Names: Sinus floor augmentation

SUMMARY:
Implant placement in posterior maxilla is often compromised or impossible due to atrophy of the bone and pneumatisation of the maxillary sinus. Thus, alveolar ridge augmentation is frequently necessary. The most commonly used method to augment the maxillary region involves the maxillary sinus floor augmentation (MSFA) with autogenous bone graft or bone substitute. Harvesting of autogenous bone graft is associated with risk of donor site morbidity and unpredictable resorption of the graft. Thus, bone substitutes alone or in combination with autogenous bone are used increasingly.

Symbios xenograft granules is a new porcine bone mineral. Long-term studies have demonstrated that xenograft contains osteoconductive properties and is a safe grafting material. MSFA with xenograft alone or in combination with autogenous bone have shown high implant survival with new bone formation. In contrast, the maxillary sinus cavities possess significant potential for bone regeneration without the use of additional bone grafts or bone substitutes due to the principle of periosteal guided bone regeneration and surrounding bony walls. Bone regeneration after maxillary sinus membrane elevation with the use of coagulum as grafting material has shown high implant survival with new bone formation, as documented in reviews and short-term studies.

The objective is to test the H0-hypothesis of no difference in the long-term implant outcome after MSFA with 1:1 mixture of autogenous bone graft and Symbios xenograft (control) compared with the coagulum (test). Forty consecutively healthy patients with a missing posterior maxillary tooth will be allocated to test or control. Implants will be inserted simultaneously with the MSFA. Clinical and/or radiographical evaluation using periapical radiographs and Cone Beam Computer Tomography (CBCT) will be performed preoperatively, immediate postoperatively, before abutment connection, after prosthetic rehabilitation, and one year after loading to assess the implant treatment outcome and the volumetric changes of the augmented area. The primary outcome will include survival of suprastructures, survival of implants, volumetric stability of the augmented area, peri-implant marginal bone level, oral health related quality of life, and complications related to the two treatment modalities.

DETAILED DESCRIPTION:
Maxillary sinus floor augmentation (MSFA) is used to enhance the alveolar bone height of the posterior maxilla. Autogenous bone is the preferred graft material. Dental implants inserted in sinuses augmented with autogenous bone grafts have demonstrated high implant survival. However, autogenous bone grafts is associated with risk of donor site morbidity and unpredictable graft resorption. Hence, various bone substitutes alone or in combination with autogenous bone graft are used to simplify the surgical procedure by diminishing the need for bone harvesting. Reviews have reported high survival of suprastructures and implants after MSFA with different mixtures of autogenous bone graft and bone substitutes. Xenograft is a tissue graft transplanted from another species than humans. MSFA with xenograft alone or in combination with autogenous bone graft have demonstrated high survival of suprastructures and implants. Symbios xenograft granules (Dentsply, United Kingdom) is a new porcine bone mineral characterized as an anorganic bone matrix with an interconnecting pore structure that supports formation and in-growth of new bone. A short-term study comparing autogenous bone graft with porcine bone alone or a mixture of autogenous bone and porcine bone indicated that porcine bone alone or in combination with autologous bone is biocompatible and osteoconductive and can be successfully used for MSFA. However, the long-term implant survival after MSFA with autogenous bone graft in combination with Symbios xenograft granules is presently unknown. In contrast, it has been postulated that bone formation in the maxillary sinus does not require the presence of a grafting material. The maintenance of space for blood clot formation accompanied by the resorption and deposition of bone cells derived from the sinus periosteum or cancellous bone of the maxilla would be responsible for bone formation. Moreover, high implant survival rate, limited peri-implant marginal bone loss, few biological and technical complications has been documented after MSFA with blood coagulum as grafting material. However, only few short-term studies have compared MSFA with blood coagulum and autogenous bone graft or bone substitutes. Therefore, it is presently unknown how much bone regeneration and grafting is necessary for long-term functional implant stability after MSFA.

Purpose Test the H0-hypothesis of no difference in implant treatment outcome after MSFA with a 1:1 mixture of autogenous bone graft and Symbios xenograft granules compared with blood coagulum as grafting material. Assessment will include survival of suprastructures and implants, changes in peri-implant marginal bone level, volumetrical stability of the graft material and treatment related complications after an observation period of one year. Oral health related quality of life (OHIP-14) and patient satisfaction will also be assessed using questionnaire and visual analogue scales (VAS).

Objective

Test the H0 hypothesis of no differences in:

* Survival of suprastructures and implants.
* Volumetrical stability of the graft.
* Peri-implant marginal bone level.
* Implantat stability quotient.
* Patient-reported outcome measures.
* Complications.

Outcome measures

Primary outcome measures:

* Survival of suprastructures. Loss of suprastructures is defined as a total loss because of a non-treatable mechanical/or biological complication.
* Survival of implants. Loss of implants is defined as removal of a non-integrated implant, mobility of previously clinical osseointegrated implant, and removal of non-mobile implants due to progressive peri-implant marginal bone loss and infection.

Secondary outcome measures:

* Volumetric changes of the graft.
* Peri-implant marginal bone level.
* Patient-reported outcome measures.
* Complications e.g. loosening of crown and fractures of veneer ceramic.

Materials and methods Forty consecutively healthy patients with a missing posterior maxillary tooth will be included and randomly allocated to: 1) MSFA with a 1:1 mixture of autogenous bone graft and Symbios xenograft granules (control group) or 2) blood coagulum (test group). Patients will be included using a Facebook posting through the University's Facebook page, the local dental association website or patients that are referred to the Department of Oral and Maxillofacial Surgery, Aalborg University Hospital for treatment of a missing tooth in the posterior maxilla. All patients will be offered participation in the study, if they meet the inclusion criteria. Prior to patients' first visit, they will receive a notice informing about their rights to have a person of their choice to be present during the visit for consultation if they wish. When the patients arrive for their first visit they will be given verbal information about the study and the written information given prior to their first visit will be elaborated. They will also receive an informed consent form. Finally, patients will be informed that they are free to terminate their participation in the study at any given time without any explanation and it will not affect their further treatment.

CBCT is frequently used before and after installation of implants in conjunction with MSFA. Included patients will receive an increased radiation dose, since CBCT scanning in addition to enoral radiographs are obtained to compare the treatment modalities. Seven CBCT with a total dose of 0.609 mSV, one orthopantomogram with a dose of 0.021 mSV and seven enoral radiographs with a total dose of 0.056 mSV will be obtained and the total effective dose will be 0.686 mSV. The standard radiation dose for MSFA with a similar observation period would be 0.251 mSV. Patients participating in the study will therefore receive a higher radiation dose of 0.435 mSV compared to a standard treatment. The extra radiation that each patient in the study is exposed to equals 1 month of background radiation. The risk of getting cancer caused by radiation is 0.005% per 1 mSV. The study will include a total of 40 patients; each patient will receive an extra dose of 0.435 mSV in comparison to patients not participating in this study.

The initial examination of the patient will include:

* Clinical examination and screening.
* Missing one posterior maxillary tooth (>4 months).
* Need of one implant in the posterior maxilla.
* Adjacent tooth in opposite jaw in contact with planned crown.
* Plaque and gingival index, probing pocket depth, and probing attachment level of the adjacent tooth/teeth.
* Radiographical examination of the residual alveolar bone based on CBCT.
* Orthopantomography to document the pre-treatment status.
* Patient will fill out the OHIP-14 questionnaire. The surgical procedure will be performed in local anesthesia with or without oral sedation or in general anesthesia with nasotracheal intubation. Implant installation and fabrication of the subsequently prosthetic solution will be performed according to manufacturer's recommendations. The maxillary sinus wall is exposed by an intraoral marginal incision from tuber maxillae to the first premolar with a vertical releasing incision. A 1 x 1 cm bony window to the maxillary sinus is created with burs maintaining an intact Schneiderian membrane. The membrane is elevated from the sinus floor as well as the lateral sinus wall and displaced dorsocranially with blunt dissector. An implant bed is successively prepared on the top of the alveolar crest following manufactory's recommendations. A straight dental implant is inserted with a cover screw. The implant stability quotient is measured for all inserted implants. A sealed randomization envelope is opened in order to allocate the patient to: 1) 1:1 mixture of autogenous bone graft and Symbios xenograft granules or 2) blood coagulum. The autogenous bone graft is harvested with a curved SafeScraper from the zygomatic buttress. Specially prepared stainless steel cup are used to estimate 1 cm3 of particulated autogenous bone graft, which will be mixed with 1 ml of Symbios xenograft granules (0.25-1 mm) and soaked in autogenous blood until use. Approximately two ml blood coagulum will be sucked from the surgical area. In the control group, the sinus around the implant is packed with the 1:1 mixture of autogenous bone graft and Symbios xenograft granules. In the test group, the sinus around the implant is filled with a two ml blood coagulum around the inserted implant. Periosteum and mucosa are sutured with Vicryl 4-0. No provisional restoration is inserted during the healing period. Patient questionnaire will be filled out after one week and one month. After six months of healing, inserted implants are exposed via a crestal incision and implant stability quotient is measured before healing abutment is placed. Mucosa is adapted and sutured with Vicryl 4-0. The prosthetic restoration will be initiated three weeks after the healing abutment has been placed including individualized abutment and fixed restoration.

Patients will be scheduled for a postoperative clinical examination after one year of loading involving:

* Plaque and gingival index, probing pocket depth, and probing attachment level.
* Oral health related quality of life - OHIP-14.
* Patient satisfaction (VAS). Oral Health Impact Profile (OHIP) is a questionnaire designed to measure impairment of oral health related quality of life and focuses on the frequency of complaints regarding the general dentition over a course of time. However, OHIP states the patient's overall oral impairment, and does not take a specific treatment site into account. Therefore, additional questionnaire including VAS may be used to evaluate the area of a missing tooth and/or a tooth replacement. The total implant treatment, peri-implant soft tissues, implant crown, and implant function at the follow-up examination will be assessed using a systematic questionnaire. Each question will be scored on a 100-mm VAS with 0 indicating extreme dissatisfaction and 100 indicating complete satisfaction. The VAS scores will be measured to the nearest mm by a ruler.

Radiographical evaluation will include seven sets of periapical radiographs and CBCT-scan obtained preoperatively, immediately postoperatively, after abutment connection and after 1 year of loading. To provide blinding of the radiographical evaluation, the CBCT-scans are coded. Volumetrical changes of the grafts are estimated by point counting and the method described originally by Cavalieri. To obtain an equivalent starting point for the systematic uniform random sampling of the CBCT-scans images involving the maxillary sinus, all images from the neighboring teeth to the implant bed are selected. The first CBCT images after the distal surface of the anterior neighboring tooth is sampled randomly using a random number table for each maxillary sinus. Every second CBCT image is selected to ensure an equal mutual distance between the selected 5-10 images. The original outline of the maxillary sinus before implant installation is recorded and superimposed on the corresponding images. A point grid test system is superimposed at random on all images, allowing 100-200 points to hit the graft of each maxillary sinus. The numbers of intersections over the graft are counted on each selected image. Cavalieri volume estimation principle is used to estimate the total volume of the graft.

Peri-implant marginal bone changes are evaluated by linear measurements on digital periapical radiographs at implant placement, baseline and one year after loading. The distance from the implant-abutment connection to the marginal bone level will be measured mesially and distally parallel with the long-axis of the implant.

ELIGIBILITY:
Inclusion Criteria:

* ≥20 years.
* Missing one posterior maxillary tooth.
* Residual bone height of the maxillary alveolar process ≥4-7 mm≤.
* Width of the alveolar process ≥6.5 mm.
* Mandibular occluding teeth.

Exclusion Criteria:

* Contraindications to implant therapy.
* Full mouth plaque score >25%.
* Progressive marginal periodontitis.
* Acute infection in the area intended for implant placement.
* Parafunction, bruxism, or clenching.
* Psychiatric problems or unrealistic expectations.
* Heavy tobacco use, define as >10 cigarettes per day.
* Pregnancy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival of suprastructures | After one year of functional loading
  Loss of suprastructures is defined as a total loss because of a non-treatable mechanical/or biological complication
Survival of implants | After one year of functional loading
  Loss of implants is defined as removal of a non-integrated implant, mobility of previously clinical osseointegrated implant, and removal of non-mobile implants due to progressive peri-implant marginal bone loss and infection

SECONDARY OUTCOMES:
Volumetric changes of the graft material | One year after sinus floor elevation and augmentation
  Estimated by CT-scan
Peri-implant marginal bone level | One year of functional loading
  Estimated by x-ray

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University Hospital, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No
Patient data will not be shared